CLINICAL TRIAL: NCT00317239
Title: Comparison of Safety & Efficacy of a Unique Intravenous Iron (VIT45) Preparation vs Oral Iron in the Treatment of Anemia in Non-Dialysis Dependent Chronic Kidney Disease
Brief Title: VIT45 Versus Oral Iron in the Treatment of Anemia in Non-Dialysis Dependent Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT04004
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: Anemia; Chronic Kidney Disease; Iron
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Iron-Dextran Complex; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): A maximum dose of 1,000 mg of FCM over 15 minutes on day 0, and a maximum dose of 500 mg of FCM over 15 minutes on days 17 and 31 based on Ferritin and TSAT values.
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Ferrous Sulfate tablets (Active Comparator): 325 mg/TID x 8 weeks
  Interventions: Drug: Ferrous Sulfate tablets

INTERVENTIONS:
Drug: Ferrous Sulfate tablets — 325 mg/TID x 8 weeks
  Arms: Ferrous Sulfate tablets
Drug: Ferric Carboxymaltose (FCM) — A maximum dose of 1,000 mg of FCM over 15 minutes on day 0, and a maximum dose of 500 mg of FCM over 15 minutes on days 17 and 31 based on Ferritin and TSAT values.
  Arms: Ferric Carboxymaltose (FCM)

SUMMARY:
This study compares the efficacy and safety of intravenous (IV) iron (VIT45) versus oral iron (ferrous sulfate) administered to subjects who suffer from anemia and are diagnosed with non-dialysis dependent chronic kidney disease (NDD-CKD).

DETAILED DESCRIPTION:
This study compares the efficacy and safety of intravenous (IV) iron (VIT45) versus oral iron (ferrous sulfate) administered to subjects who suffer from anemia and are diagnosed with non-dialysis dependent chronic kidney disease (NDD-CKD).

ELIGIBILITY:
Inclusion Criteria:

* Males or females > or = 12 years of age
* NDD-CKD subjects
* Baseline hemoglobin < or = 11g/dl
* Stable erythropoietin (EPO) status

Exclusion Criteria:

* Known hypersensitivity to ferrous sulfate or IV iron
* Unstable EPO status
* Anemia not related to CKD
* Chronic, serious infection
* Recent IV iron
* Recent blood transfusion
* Recent blood loss
* Need for surgery
* Received investigational drug within 30 days
* Female subjects who are pregnant or lactating

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

REFERENCES:
- [Result] Qunibi WY, Martinez C, Smith M, Benjamin J, Mangione A, Roger SD. A randomized controlled trial comparing intravenous ferric carboxymaltose with oral iron for treatment of iron deficiency anaemia of non-dialysis-dependent chronic kidney disease patients. Nephrol Dial Transplant. 2011 May;26(5):1599-607. doi: 10.1093/ndt/gfq613. Epub 2010 Oct 7. PMID 20929915
- [Result] Qunibi W, Martinez C, Smith M, Benjamin J, Dinh Q. A Randomized Controlled Trial Comparing IV Ferric Carboxymaltose (FCM) to Oral Iron in Anemic Patients with Non-Dialysis-Dependent CKD. American Society of Nephrology Renal Week 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets
Started | 147 | 103
Completed | 134 | 84
Not Completed | 13 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets | Total
Number analyzed (Participants) | 147 | 103 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 42 | 107
  >=65 years | 82 | 61 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (12.56) | 66.8 (13.48) | 65.94 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 73 | 167
  Male | 53 | 30 | 83
Region of Enrollment [Number; unit: participants]
  United States | 147 | 103 | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving an Increase in Hemoglobin ≥1g/dL
Time Frame: anytime during the study
Population: Modified Intent to Treat (mITT) population defined as subjects who received at least 1 dose of study medication, had stable EPO for at least 8 weeks prior to randomization, had at least 1 post-baseline hemoglobin assessment, and who had NDD-CKD characterized by a GFR ≤45 mL/min/1.73²
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets
Number analyzed (Participants) | 144 | 101
participants | 87 | 35

ADVERSE EVENTS:
Time Frame: 1 year and 9 months
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets
Serious Adverse Events (participants affected / at risk) | 13/147 | 10/103
Other Adverse Events (participants affected / at risk) | 11/147 | 20/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=147) | Ferrous Sulfate Tablets (N=103)
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=147) | Ferrous Sulfate Tablets (N=103)
Constipation (Gastrointestinal disorders) | 2 | 18
Odema peripheral (General disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less